CLINICAL TRIAL: NCT05489666
Title: Effects of Vitamin D on Skeletal Muscle Strength in Resistance Trained Adult Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Nilophar Zandieh, MS, Principle Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-306
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Nutrition Status; Nutritional Requirements; Sports Nutritional Sciences
Keywords: Nutrition; Supplement; Supplementation; Vitamin D; Strength Training; Resistance Training; Women; Female; Athlete

STUDY DESIGN:
Intervention Model Description: A two-arm parallel assignment; one group receives the treatment (vitamin D3 supplement 5,000IU/day) and one group receives the placebo (control).
Who Masked: Participant, Investigator
Masking Description: Double-blind masking; neither the investigator nor the participants will know, the assigned intervention placement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Active Comparator): Participants in this group will be administered an oral Vitamin D3 supplement; 5,000 IU/ day. The participants will take the supplement themselves, orally, once per day, for 8 weeks.
  Interventions: Dietary Supplement: Nature Made Vitamin D3 5,000 IU, 125mcg
- Control Group (Placebo Comparator): Participants in this group will be administered an oral, soft-gel, lookalike placebo. The participants will take the supplement themselves, orally, once per day, for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nature Made Vitamin D3 5,000 IU, 125mcg — Taking a 5,000 IU oral supplement of Vitamin D3, daily, for 8 weeks, may improve strength performance in women who have and are continuing a resistance trained workout regimen. After blood vitamin D levels have been raised to an optimal range, a lower dosage may be assigned as needed from 5,000 IU per day to 1,000-2,000 IU per day.
  Other Names: Spring Valley; Life Extensions; GNC; Nature's Bounty; CVSHealth; Swanson
  Arms: Treatment Group
Dietary Supplement: Placebo — Resistance trained women may not improve their strength performance with low levels of vitamin D in the blood.
  Arms: Control Group

SUMMARY:
The majority of vitamin D research has been done in non-athletic populations, particularly older populations, to analyze muscle weakness, pain, balance, and fractures. It has been reported that over a billion people worldwide are vitamin D deficient, including 36-70% of the young adult population. Previous literature also suggests that, even among healthy athletes, over 50% of subjects sampled had inadequate or insufficient vitamin D levels. Vitamin D deficiency can occur in young women, including pregnant women, and the risk of deficiency is even higher with advancing age in a woman's lifecycle. It is known that preserving skeletal muscle (SM) function is critical for women of all ages to prevent sarcopenia. Two factors in preserving SM are protein intake and resistance training. Relatively unknown are the actions of Vitamin D on SM function. Vitamin D deficiency can have a negative effect on SM function . However, additional research is needed to investigate the increase in SM strength when the serum concentration of vitamin D is improved. It is possible that an athlete may require an increased intake of vitamin D to assure adequate availability and storage for optimal performance; however, is known that food sources of vitamin D are limited in sufficient quantity to meet these requirements. Athletes who are insufficient will require a supplement of vitamin D3 for up to 5000 IU/day for at least eight weeks, to potentially reach optimal levels, then 1000-2000 IU/day for maintenance.

DETAILED DESCRIPTION:
The investigators seek to determine if women with a vitamin D serum concentration lower than 50 nmol/L and who regularly resistance train will improve strength performance outcomes when taking a daily supplement of 5000 IU of vitamin D3 over an 8-week period, as compared to the same demographic of women who do not take a daily supplement of vitamin D3. The participants will receive "Nature's Bounty Vitamin D3, 5,000 IU, soft gels" and the PI will be providing the supplement and the placebo. A pre-intervention data collection and screening (PRE) will be performed involving blood draw, food log, a body composition test (using Dual-energy X-ray absorptiometry [DEXA]), and a BioDex testing to determine maximal muscle strength. Following PRE testing, the participants will be divided into one of two groups: 1) taking a vitamin D3 supplement (n=20) or, 2) taking a placebo. The participants will be instructed to continue their resistance training regimen. Training will be logged and turned in to the PI weekly. The participants will perform a post-intervention data collection (POST), which includes the same test from PRE. Variables of interest will include changes in: 1) blood level of vitamin D, 2) muscle and fat mass, and 3) leg strength/power during the BioDex test.

ELIGIBILITY:
Inclusion criteria will include:

Participant will need to answer "yes" to the following items:

1. female
2. not pregnant
3. between the ages of 19-55 years old
4. a non-smoker
5. currently resistance training (i.e., lifting weights) for more than 2 days/week for a minimum of > 24 months
6. free of any known overt cardiovascular or metabolic disease
7. not an active user of tanning beds
8. not consuming now or haven't consumed within the last 6 months, a vitamin D or multivitamin supplement or a form of a supplement with vitamin D added
9. not consuming now or haven't consumed within the last 2 months, agents that affect hormones (testosterone boosters, growth hormone boosters, etc.) (does not include birth control/oral contraceptives)
10. not allergic to rubbing alcohol

Exclusion criteria will include:

1) Outside of study inclusion parameters

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Biodex Strength performance change | 8 weeks
  Taking a daily supplement of 5,000 IU of vitamin D3 may change strength outcomes measured in newton meters (Nm).

SECONDARY OUTCOMES:
Serum 25(OH)D status | 8 weeks
  Taking a daily supplement of 5,000 IU of vitamin D3 may change blood levels of vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Donna O Burnett, PhD, Study Chair — Auburn University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams GD, Feldman D, Safran MR. Effects of Vitamin D on Skeletal Muscle and Athletic Performance. J Am Acad Orthop Surg. 2018 Apr 15;26(8):278-285. doi: 10.5435/JAAOS-D-16-00464. PMID 29561306
- [Result] Bartoszewska M, Kamboj M, Patel DR. Vitamin D, muscle function, and exercise performance. Pediatr Clin North Am. 2010 Jun;57(3):849-61. doi: 10.1016/j.pcl.2010.03.008. PMID 20538161
- [Result] Chiang CM, Ismaeel A, Griffis RB, Weems S. Effects of Vitamin D Supplementation on Muscle Strength in Athletes: A Systematic Review. J Strength Cond Res. 2017 Feb;31(2):566-574. doi: 10.1519/JSC.0000000000001518. PMID 27379960
- [Result] Dahlquist DT, Dieter BP, Koehle MS. Plausible ergogenic effects of vitamin D on athletic performance and recovery. J Int Soc Sports Nutr. 2015 Aug 19;12:33. doi: 10.1186/s12970-015-0093-8. eCollection 2015. PMID 26288575
- [Result] Han Q, Li X, Tan Q, Shao J, Yi M. Effects of vitamin D3 supplementation on serum 25(OH)D concentration and strength in athletes: a systematic review and meta-analysis of randomized controlled trials. J Int Soc Sports Nutr. 2019 Nov 26;16(1):55. doi: 10.1186/s12970-019-0323-6. PMID 31771586
- [Result] Knechtle B, Nikolaidis PT. Vitamin D and Sport Performance. Nutrients. 2020 Mar 21;12(3):841. doi: 10.3390/nu12030841. PMID 32245151
- [Result] Ksiazek A, Zagrodna A, Slowinska-Lisowska M. Vitamin D, Skeletal Muscle Function and Athletic Performance in Athletes-A Narrative Review. Nutrients. 2019 Aug 4;11(8):1800. doi: 10.3390/nu11081800. PMID 31382666
- [Result] Ogan D, Pritchett K. Vitamin D and the athlete: risks, recommendations, and benefits. Nutrients. 2013 May 28;5(6):1856-68. doi: 10.3390/nu5061856. PMID 23760056
- [Result] Stockton KA, Mengersen K, Paratz JD, Kandiah D, Bennell KL. Effect of vitamin D supplementation on muscle strength: a systematic review and meta-analysis. Osteoporos Int. 2011 Mar;22(3):859-71. doi: 10.1007/s00198-010-1407-y. Epub 2010 Oct 6. PMID 20924748
- [Result] Tomlinson PB, Joseph C, Angioi M. Effects of vitamin D supplementation on upper and lower body muscle strength levels in healthy individuals. A systematic review with meta-analysis. J Sci Med Sport. 2015 Sep;18(5):575-80. doi: 10.1016/j.jsams.2014.07.022. Epub 2014 Aug 11. PMID 25156880
- [Result] Wicinski M, Adamkiewicz D, Adamkiewicz M, Sniegocki M, Podhorecka M, Szychta P, Malinowski B. Impact of Vitamin D on Physical Efficiency and Exercise Performance-A Review. Nutrients. 2019 Nov 19;11(11):2826. doi: 10.3390/nu11112826. PMID 31752277
- [Result] de la Puente Yague M, Collado Yurrita L, Ciudad Cabanas MJ, Cuadrado Cenzual MA. Role of Vitamin D in Athletes and Their Performance: Current Concepts and New Trends. Nutrients. 2020 Feb 23;12(2):579. doi: 10.3390/nu12020579. PMID 32102188